CLINICAL TRIAL: NCT02660099
Title: Internet Delivered Cognitive Behavior Therapy for Obsessive-compulsive Disorder in Adolescents With Autism Spectrum Disorder - A Clinical Case Series
Brief Title: Internet Delivered CBT for OCD in Adolescents With ASD - A Clinical Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Serlachius, Research director, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BiP-ASD/OCD
Record Dates: First submitted 2015-07-07; First posted 2016-01-21 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Obsessive Compulsive Disorder; Autism Spectrum Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet-delivered CBT (Experimental): 12 weeks of internet-delivered cognitive behavior therapy provided through a secure internet platform and online clinician contact
  Interventions: Behavioral: Internet-delivered Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavior Therapy — The treatment consists of standard cognitive behavior therapy for obsessive-compulsive disorder and is delivered via an internet platform and regular therapist contact several times per week via email and telephone. The treatment is 12 weeks. Both parents and adolescents are involved in treatment. Parents will also receive three lectures on 1, Autism spectrum disorder, 2, CBT and functional analysis and 3, Parental strategies

SUMMARY:
The aim of this study is to test the feasibility and acceptability of an internet-delivered cognitive behavior therapy (ICBT) intervention originally developed for neurotypical adolescents with obsessive compulsive disorder (OCD) in adolescents with OCD and autism spectrum disorder (ASD). This feasibility study will inform us how to adapt the original intervention to the specific needs of patients with ASD.

DETAILED DESCRIPTION:
To evaluate the effectiveness of ICBT for OCD in adolescents with ASD, this study will use a single case experimental design with weekly measures during two phases: A-B. The A-phase will consist of baseline measures at least three weeks prior to treatment. The B-phase will consist of the 12 weeks ICBT-program as well as one measure post-treatment. Single case descriptions of each participant will be presented. Weekly measures on the Obsessional Compulsive Inventory - Child version (OCI-CV) will be analyzed through visual inspection of each participants graph and through computation of Percentage of Non-overlapping Data (PND). PND is a frequently used effect measure in SCED and reflects how large percentage of the measurements during the treatment-phase that do not overlap with any of the measurements during the base-line phase.

To assess the feasibility and comprehension of the ICBT treatment semi-structured interviews (face-to-face or telephone) will be conducted with participants and parents weekly during the four first weeks of ICBT and semi-weekly during the rest of the treatment. Detailed notes will be taken during each interview and will serve as content material for a thematic analysis trying to determine possible accommodations to the ICBT protocol to better suit patients with ASD.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of OCD as defined by DSM-5 [40]
* a diagnosis of autism defined by DSM-5
* a total score of ≥ 16 on the Children's Yale-Brown Obsessive-Compulsive Scale, CY-BOCS [14]
* age between 12 and 17 years
* ability to read and write Swedish
* access to the internet
* a parent that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* psychosis or bipolar disorder, severe eating disorder
* suicidal ideation
* subject not able to read or understand the basics of the ICBT material
* completed CBT for OCD within last 12 months (defined as at least 5 sessions of CBT including exposure and response prevention)
* ongoing psychological treatment for OCD or another anxiety disorder

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Obsessional Compulsive Inventory - Child version, OCI-CV | Change from baseline to 12 weeks
  Self-rated OCD symptom levels

SECONDARY OUTCOMES:
Children's Yale Brown Obsessive Compulsive Scale | Change from baseline to 12 weeks
  Clinician-rated OCD symptom levels
Mini International Neuropsychiatric Interview for Children and Adolescents, MINI-KID | Baseline
  psychiatric screening of comorbidity
Clinical Global Impression - Severity, CGI-S | Change from baseline to 12 weeks
  Global symptom levels
Clinical Global Impression - Improvement, CGI-I | Post treatment(12 weeks)
  Global symptom improvement
Children's Global Assessment Scale, CGAS | Change from baseline to 12 weeks
  Global level of functioning
Children´s Depression Inventory - Short version | Change from baseline to 12 weeks
  Symptom level of depressive mood
Strength and difficulties, SDQ | Change from baseline to 12 weeks
  General psychopathology
Family Accommodation Scale, Parent-Report, FAS-PR | Change from baseline to 12 weeks
  Parental accommodation to OCD symptoms
Patient ICBT Adherence Rating, PIAR | after 6 weeks and at post treatment(12 weeks)
  Patient Adherence to internet delivered CBT
Education, Work and Social Adjustment Scale - child and parent version, EWSAS | Change from baseline to 12 weeks
  Global functioning

CONTACTS AND LOCATIONS:
Overall Officials: David Mataix-Cols, Professor, Principal Investigator — Department of Clinical Neuroscience, Karolinska Institutet
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Karolinska insititute, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided